CLINICAL TRIAL: NCT04024475
Title: Prospective Cohort Study With Collection of Clinical Data, Serum and Plasma of Patients With Prostate Disease
Brief Title: Prostate Cancer Biobank
Status: Active, not recruiting | Type: Observational
Sponsor: Swiss Cancer Institute (Other)
Collaborators: ProteoMediX AG (Industry); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Other Study IDs: SAKK 63/12
Record Dates: First submitted 2019-07-11; First posted 2019-07-18 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Prostatic Neoplasms
Keywords: Radical prostatectomy; Metastatic castration resistant prostate cancer; Oligometastatic prostate cancer; Radiotherapy; Prostate cancer screening; Prostate-specific antigen (PSA); Prostate cancer (PCa); Opportunistic screening
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Serum, plasma, and buffy coat samples; Prostate biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- A: Opportunistic screening & benign prostate syndrome (BPS): Asymptomatic men offered screening (PSA testing) with prostate biopsy (A1). Or patients with lower urinary tract symptoms from benign prostatic hyperplasia undergoing: no treatment (A2), medical therapy (A3), or transurethral resection of the prostate (A4)
  Interventions: Other: Observation
- B: Localized/locally advanced PCa with curative intent: B0: Patients under active surveillance (B0, closed group); B1: radical prostatectomy (RP) or RP followed by (adjuvant) external beam radiation; B2: external beam radiation therapy (EBRT) without androgen deprivation therapy (ADT); B3: external beam radiation therapy with ADT
  Interventions: Other: Observation
- C: Biochemical relapse: Patients with PSA progression after RP with or without systemic therapy
  Interventions: Other: Observation
- D: Metastatic PCa but hormone sensitive: Metastatic PCa without curative treatment but hormone sensitive disease, treated with ADT (medical or surgical), with or without additive treatments. Oligometastatic PCa.
  Interventions: Other: Observation
- E: Metastatic castration resistant prostate cancer (mCRPC): Metastatic castration resistant prostate cancer (mCRPC). Oligometastatic PCa.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
Carcinoma of the prostate is the second most commonly diagnosed cancer and occurs predominantly in older men - almost two-thirds of those affected are over 65 years of age. In a significant proportion of patients, the disease is harmless and progresses only very slowly. As a result, there is a risk of overdiagnosis and overtreatment. The main diagnostic tool for prostate cancer is the prostate-specific antigen (PSA) test, but its specificity is minimal. It is important to look for other biological characteristics (biomarkers) that provide pointers to the need for a diagnosis and treatment. Even after treatment and in advanced stages of disease, decisions are often difficult, because it is not necessarily clear which patient needs a specific treatment.

In this study, a multicenter biobank of patient sera, plasma and tissue is being established together with information of relevance to the disease, in order to provide a basis for the testing of biomarkers. The aim is to identify markers that offer diagnostic and treatment-selective pointers and thus make a decisive contribution to the optimum care of patients.

DETAILED DESCRIPTION:
Background & Rationale:

Prostate Cancer (PCa) occurs mainly in older men, nearly two thirds are diagnosed in men aged 65 or older. However, in a substantial subset of patients, the disease will be slow-growing and harmless. This highlights one of the major issues with PCa screening and diagnosis: the risks of over-detection and overtreatment, i.e. to diagnose and invasively treat indolent cancers that may lead to reduced quality of life without increasing overall survival.

The main diagnostic tool for PCa is the systematic screening for PSA (prostate-specific antigen), despite the low specificity of PSA and the unclear cut-off value, resulting in a large proportion of unnecessary biopsies with potential side effects. Additionally, as screening addresses a healthy population and screened men may suffer from disadvantages, such as unnecessary biopsies, screening in PCa remains controversial.

Besides the dilemmas in PCa screening, there are several additional important clinical questions that deserve further investigation and better risk-adapted patient stratification as follows: 1) active treatment versus deferred therapy in the heterogeneous group of patients with localized PCa; 2) treatment intensification for locally-advanced, high-risk prostate cancers with significant risk of PCa-related deaths; 3) optimal approach for patients with high risk of local recurrence post-radical prostatectomy; 4) treatment of patients with rising PSA (biochemical relapse) after curative treatment (either radical prostatectomy or RT); 5) a better understanding of oligometastatic disease and; and 6) treatment of patients with castration-resistant prostate cancer (CRPC).

PCa is characterized by a wide spectrum of molecular and phenotypic characteristics. PCa patients are currently grouped in different risk categories, illustrating particular features of a heterogeneous disease. On one side, many patients present benign disease, such as benign prostate enlargement caused by prostate hyperplasia and, on the other side, progressively malignant PCa, ranging from localized, locally-advanced, metastatic and castrate-resistant disease.

For the purpose of this study, we established 5 groups and their corresponding subgroups, as follows:

A) Opportunistic screening and benign prostate syndrome (BPS) with prostate biopsy; B) Localized and locally advanced prostate cancers treated with curative intent; C) Biochemical relapse after RP; D) Metastatic advanced PCa without curative treatment but hormone sensitive disease, treated with ADT (medical or surgical); E) Metastatic castration resistant prostate cancer (mCRPC).

Currently a comprehensive biobank in the field of urogenital disease, driven by a multidisciplinary panel (composed by specialists from the following fields: urology, medical oncology, radio-oncology and pathology), does not exist in Switzerland.

Such biobank (together with the corresponding clinical data) would enable researchers and clinicians alike to discover and validate diagnostic, prognostic and predictive PCa biomarkers, which are currently highly needed.

Importantly, the biobank shall consist of specific sample sets related to the different stages of PCa development (including screened healthy men and newly diagnosed patients). Ultimately, this comprehensive project will allow addressing some of the urgent questions in different stages of PCa.

Objective:

To create a novel and comprehensive plasma and serum biobank of about 55000 samples (derived from about 1540 patients) accompanied by the corresponding clinical data. This will enable us to explore and validate different diagnostic, prognostic and predictive biomarkers regarding prostate disease.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for storage of liquid samples and referencing of biopsy(-ies) in the biobank, and for clinicopathological data collection, for translational research purposes.

Criteria for entering diagnostic group A

* Patient scheduled for prostate biopsy for any reason

Criteria for entering group B

Subgroup B0 (active surveillance, closed group):

* Patient under active surveillance for localized PCa

All of the following criteria should be fulfilled:

* clinical stage T1/T2
* PSA ≤ 10 ng/ml
* PSA density < 0.2 ng/ml per milliliter
* biopsy Gleason score ≤ 6
* one or two positive biopsy cores

Subgroups B1-B3 (treatment with curative intent):

* Patient under treatment for localized PCa with either radical prostatectomy or RP followed by (adjuvant) external beam radiation (B1), or external beam radiation therapy without (B2) or with ADT (B3).

Criteria for entering diagnostic group C

* Patient underwent RP
* Patient with biochemical relapse: PSA progression after RP is defined as two consecutive rises with final PSA value > 0.1 ng/mL, or three consecutive rises (the first value must be measured earliest 4 weeks after radical prostatectomy).
* Patient is candidate for salvage RT with or without combined systemic therapy.

Criteria for entering diagnostic group D

* Metastatic PCa without curatively intended treatment, but hormone sensitive disease, treated with ADT (medical or surgical) with or without additive treatments, such as docetaxel or short term course of Bicalutamide or continuous Bicalutamide.
* Oligometastatic PCa: N1 or M1a/b disease detected on PET or whole body MRI presenting ≤5 synchronous lesions (bone and/or lymph nodes), under active surveillance, or treated with chemotherapy, treated with focal RT (i.e. SBRT), treated with surgery or other treatments; ADT can be combined, but it is not necessarily required for oligometastatic patients.

Criteria for entering diagnostic group E (metastatic castration resistant PCa)

* Patient with mCRPC defined by: progressive disease after surgical castration or under medical ADT and suppressed testosterone levels.
* Oligometastatic PCa: N1 or M1a/b disease detected on PET or whole body MRI presenting ≤5 synchronous lesions (bone and/or lymph nodes), under active surveillance, or treated with chemotherapy, treated with focal RT (i.e. SBRT), treated with surgery or other treatments; ADT can be combined, but it is not necessarily required for oligometastatic patients.

Exclusion criteria:

* Other concurrent active malignancy.
* Psychiatric disorder precluding understanding of information on study related topics and giving informed consent.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See description under "Groups/Cohorts"
Sampling Method: Probability Sample
Enrollment: 1323 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Group A: Time to prostate cancer (PCa) histological diagnosis | At the occurrence of a positive biopsy result or latest 10 years after registration
  Time to PCa histological diagnosis will be calculated from the time when patients were assigned into group A until documentation of a positive biopsy result.
Group B0: Progression free survival (PFS) | At 1 year after assigned into Group B0
  PFS will be calculated from the time when patients were assigned into group B0 until first documented event occurred:
  * three or more positive cores at rebiopsy
  * Gleason score ≥ 7 at rebiopsy
Group B1: Biochemical relapse free survival | At 5 years after assigned into Group B1
  Biochemical relapse free survival is calculated from the time when patients were assigned into group B1 until prostate specific antigen (PSA) relapse occurs. PSA relapse is defined as PSA progression after radical prostatectomy (RP) is defined as two consecutive rises with the final PSA value > 0.1 ng/mL, or three consecutive rises (the first value must be measured earliest 4 weeks after RP).
Group B2-B3: Interval to biochemical failure (IBF) | At 18 months after assigned into Group B2-B3
  IBF is defined as the time interval from completion of treatment by patients of group B2 or B3 until biochemical failure (BF). BF is defined by an absolute PSA value superior or equal to the post-treatment PSA nadir + 2 ng/mL.
Group C: Progression free survival (PFS) | At progression or latest 10 years after assigned into Group C
  PFS is counted from the day the patient entered group C to the day of the first record of either local or regional recurrence, distant recurrence, start of hormonal treatment after biochemical failure, or death due to any cause.
Group D: Biochmical prostate specific antigen progression | At 6 months after induction of androgen deprivation therapy
  The biochemical prostate specific antigen (PSA) progression is calculated from the induction of palliative androgen deprivation therapy (ADT), defined as:
  * In case PSA levels had not decreased from baseline, under treatment: ≥ 25% increase from baseline (last PSA measurement before treatment start) AND an increase in the absolute PSA value of ≥ 2 ng/mL and presence of castrate level of testosterone.
  * In case PSA levels decreased from baseline, under treatment: ≥ 25% increase above the nadir AND an increase in the absolute PSA value of ≥ 2 ng/mL and presence of castrate level of testosterone.
Group E: Overall survival (OS) | At death or latest 10 years after assigned into Group E
  OS will be calculated from the time when patients were assigned into group E until death from any cause. OS will be censored at the time the patient is last known to be alive if:
  * the patient is lost to follow-up
  * or death is not experienced.

SECONDARY OUTCOMES:
Group A, B0-B3, C, D: Overall survival (OS) | At death from any cause or latest 10 years after assigned into the corresponding Group
  OS will be calculated from the time when patients were assigned into the group until death from any cause. OS will be censored at the time the patient is last known to be alive if:
  * the patient is lost to follow-up
  * or death is not experienced.
Group A, B1-B3, C: Time to PCa-specific death | At prostate cancer related death or latest 10 years after assigned into the corresponding Group
  Time to PCa-specific death is calculated from the time when patients were assigned into the group until death due to cancer occurs.
Group B0: Progression free survival (PFS) | At the occurrence of the event or latest 10 year after assigned into Group B0
  PFS will be calculated from the time when patients were assigned into group B0 until first documented event occurred:
  * three or more positive cores at rebiopsy
  * Gleason score ≥ 7 at rebiopsy
  * after follow-up ≥ 1 year: PSA doubling time <3 years
Group B0: Event free survival (EFS) | At the occurrence of the event or latest 10 year after assigned into Group B0
  EFS will be calculated from the time when patients were assigned into group B0 until documented events, whichever occurs first:
  * Any criteria defining PFS, and in addition the following ones:
  * transurethral resection
  * RP with curative intent
  * RT with curative intent
  * start of androgen deprivation therapy (ADT)
Group D: Progression free survival (PFS) | At the occurrence of the event or latest 10 year after assigned into Group D
  PFS is calculated from the time when patients were assigned into group D until documentation of one or any combination of the following events occurred:
  * Biochemical PSA progression
  * Progression of metastatic disease
  * symptomatic clinical progression
  * death
Group E: Progression free survival (PFS) | At the occurrence of the event or latest 10 year after assigned into Group E
  PFS will be calculated from the time when patients were assigned into group E until disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Engeler, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (12):
- Switzerland (12):
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubuenden, Chur
  - Hopital Fribourgeois HFR, Fribourg
  - Hôpitaux Universitaires Genève HUG, Geneva
  - Luzerner Kantonsspital, Lucerne
  - Clinica Luganese, Lugano
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital STS AG, Thun

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared on reasonable request, after internal and ethical approval
URL: http://sakk.ch